CLINICAL TRIAL: NCT00485537
Title: Pregnancy Outcomes With a Gonadotropin-Releasing Hormone (GnRH) Antagonist (Cetrorelix) Protocol Versus GnRH-Agonist Protocol in Ovarian Stimulation for ICSI Cycles-a Prospective Study
Brief Title: Pregnancy Outcomes With a GnRH Antagonist Protocol Versus GnRH-Agonist Protocol in ICSI Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinic and Research Center in Human Reproduction Roger Abdelmassih (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA0001
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Infertility
Keywords: GnRH antagonist; GnRH agonist; ICSI; miscarriage rate; pregnancy outcome
MeSH Terms: conditions — Infertility | interventions — Oocyte Retrieval

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: oocyte retrieval and ICSI procedure

SUMMARY:
Cycles with GnRH agonist and GnRH antagonist were compared and main outcome measures were the number of oocytes retrieved, injected and fertilized, embryos transferred, and clinical pregnancy and miscarriage rates, were analized.

DETAILED DESCRIPTION:
160 women were equally divided between a GnRH antagonist protocol (Group 1) versus a GnRH agonist protocol (Group 2) in ICSI cycles. The trial was conducted between September 2005 and December 2006. The mean age in both groups was 32 (range 22-40). The main outcome measures were the number of oocytes retrieved, injected and fertilized, embryos transferred, and clinical pregnancy and miscarriage rates.

ELIGIBILITY:
Inclusion Criteria:

* Infertility couples, absence of endometriosis (confirmed by a previous surgical procedure to investigate infertility), polycystic ovarian syndrome, FSH levels < 12 IU/l, basal levels of estradiol < 20 in the group submitted to the agonist protocol and beginning of stimulation on day 2 in group submitted to antagonist protocol, in the absence of ovarian cysts on the endovaginal ultrasound

Exclusion Criteria:

* use of exogenous LH during stimulation

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2005 (Actual)
Dates: Start 2005-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Comparative response to ICSI cycles with GnRH agosnist and cetrotide | 16 months

SECONDARY OUTCOMES:
Compare number of oocytes retrieved, injected and fertilized, embryos transferred, and clinical pregnancy and miscarriage rates in both groups | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Neme, MD,PhD, Principal Investigator — Clinic and Research Center in Human Reproduction Roger Abdelmassih
Locations (1):
- Clinica e Centro de Reprodução Humana Roger Abdelmassih, São Paulo, São Paulo, Brazil